CLINICAL TRIAL: NCT03830749
Title: A Pilot Study to Evaluate the Safety and Efficacy of Eltrombopag Plus Pulsed Dexamethasone as First Line Therapy for Subjects With Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Safety and Efficacy of Eltrombopag Plus Pulsed Dexamethasone for Subjects With Idiopathic Thrombocytopenic Purpura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHRC_ITP
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Eltrombopag Oral Tablet 25-75 mg daily for 12 weeks plus pulsed dexamethasone
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag Oral Tablet 25-75 mg daily for 12 weeks plus pulsed dexamethasone

SUMMARY:
Current first line treatments for immune thrombocytopenia (ITP) usually have transient effects and prolonged platelet response rate off therapy remains low. The aim is to evaluate whether a 12-week course of eltrombopag plus pulsed dexamethasone as first line therapy can increase the proportion of patients with prolonged response. Diagnosis of ITP is established according to the American Society of Hematology guidelines. Eligible ITP subjects have platelet counts <30×109/L or counts <50×109/L and significant bleeding symptoms (WHO bleeding scale 2 or above). Subjects must have no prior ITP treatment except platelet transfusions. Treatment consists of eltrombopag 25-75 mg daily according to platelet response for 12 weeks plus pulsed dexamethasone, 40 mg daily for 4 consecutive days every 4 weeks for 1-3 courses. The primary endpoint is prolonged response rate which was defined as the proportion of enrolled subjects maintaining platelet counts >50×109/L for more than 6 months without any ITP therapy after completion of 12-week therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated a written informed consent.
2. Adults (≥18 years) diagnosed with ITP according to the American Society for Hematology/British Committee for Standards in Haematology (ASH/BCSH) Guidelines. In addition, the peripheral blood smear should support the diagnosis of ITP with no evidence of other disease causative of thrombocytopenia (e.g., pseudo thrombocytopenia, myelofibrosis). The physical examination should be normal or at least not show signs suggestive of any disease likely to be associated with thrombocytopenia.
3. No prior ITP treatment except platelet transfusions
4. Subject has no intercurrent medical event, including evidence of any thrombosis.
5. Normal prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT), no history of hypercoagulable state.
6. The following clinical chemistries must be within the normal reference range:

   creatinine, ALT, AST, total bilirubin, total albumin and alkaline phosphatase.
7. Subject is practicing an acceptable method of contraception (documented in chart).
8. Subject is able to understand and comply with protocol requirements and instructions.

Exclusion Criteria:

1. Any clinically relevant abnormality, other than ITP, identified on the screening examination, or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another diagnosis.
2. History of active malignancy or on cancer therapy. Patients with a history of malignancy in complete remission for longer than 5 years are eligible
3. History of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism).
4. ≥ two of the following risk factors: Factor V Leiden, hormone replacement therapy, systemic contraception containing estrogen, smoking, diabetes, hypercholesterolemia, medications for hypertension or cancer.
5. Pre-existing cardiac disease (including congestive heart failure, and arrhythmia requiring treatment), or clinically significant findings on resting 12-lead ECG at screening.
6. Female subjects who are nursing or pregnant (positive serum or urine β-human chorionic gonadotrophin (β-hCG) pregnancy test) at screening or pre-dose on Day 1.
7. History of alcohol/drug abuse.
8. Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The prolonged response rate | 6 months after completion of therapy
  Defined as proportion of patients with platelet counts > 50,000/μl at 6 months after completion of therapy and free of ITP rescue therapy

SECONDARY OUTCOMES:
Time to relapse | 6 months after completion of therapy
  Defined as the interval from completion of 3 months treatment to platelet count<30,000/ul and restarting of ITP therapy including but not limited to platelet transfusion, IVIG, corticosteroids, immunosuppressive drugs, rituximab
Early response rate | 6 months after completion of therapy
  Defined as proportion of patients requiring less than 3 courses of pulsed dexamethasone to maintain platelet counts > 150,000/ul
Health related quality of life | 6 months after completion of therapy
  Assessed by SV36 HRQoL questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cheng, PhD, MD, Principal Investigator — Humanity & Health Research Centre
Locations (1):
- Humanity & Health Research Centre, Hong Kong, Hong Kong SAR, Hong Kong